CLINICAL TRIAL: NCT00883168
Title: Randomized, Double-Blind Trial of MP29-02 Nasal Spray Compared to Placebo, Azelastine Hydrochloride Nasal Spray and Fluticasone Propionate Nasal Spray in the Treatment of Patients With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP4006
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Fluticasone; MP29-02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- azelastine Hcl (Active Comparator)
  Interventions: Drug: azelastineHcl
- fluticasone propionate (Active Comparator)
  Interventions: Drug: fluticasone propionate
- azelastine Hcl /fluticasone propionate (Experimental)
  Interventions: Drug: azelastine Hcl/fluticasone propionate

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: placebo
Drug: azelastineHcl — azelastine hydrochloride 548 mg
  Other Names: astelin
  Arms: azelastine Hcl
Drug: fluticasone propionate — fluticasone propionate 200 mcg
  Arms: fluticasone propionate
Drug: azelastine Hcl/fluticasone propionate — azelastine hydrochloride 548 mcg/fluticasone propionate 200 mcg
  Other Names: MP29-02
  Arms: azelastine Hcl /fluticasone propionate

SUMMARY:
The purpose of this study is to determine if the combination of two allergy medications (formulated azelastine/fluticasone product)is more effective than placebo or either component medication alone (azelastine or fluticasone).

DETAILED DESCRIPTION:
This will be a Phase III, randomized, double-blind, placebo-controlled, parallel-group study in subjects with moderate-to-severe seasonal allergic rhinitis (SAR). The study will begin with a 7-day, single-blind, placebo lead-in period (Day -7 to Day 1). Subjects will be instructed to take placebo lead-in medication twice daily (1 spray per nostril), approximately every 12 hours. On Day 1, subjects who satisfy the symptom severity requirements and continue to meet all of the study inclusion/exclusion criteria will be randomized in a 1:1:1:1 ratio to receive 1 spray per nostril twice daily of MP29-02, azelastine hydrochloride, fluticasone propionate, or placebo nasal spray.

Efficacy will be assessed by the change from baseline in the subject-reported 12-hour reflective Total Nasal Symptom Score (TNSS). On Days 1 through 14, subjects will rate the instantaneous and reflective TNSS symptoms of sneezing, nasal congestion, runny nose, and nasal itching; the instantaneous and reflective total ocular symptom score (TOSS) symptoms of itchy eyes, watery eyes and eye redness; the symptom of postnasal drip will be reflectively, twice daily (AM and PM) in a diary prior to the dose of study medication. Symptoms will be scored on a 0 to 3 scale (0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms), such that the maximum daily symptom severity score will be 24 for the TNSS and 18 for the TOSS. Additional secondary efficacy variables will include reflective individual nasal and ocular symptom scores, as well as change from Baseline to Day 14 in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ).

Subjects ≥ 18 years of age will complete the RQLQ on Day 1 (prior to dosing) and Day 14. Subjects will return to the clinic on Day 7 for an interim evaluation. After completing the 2-week double-blind treatment period, subjects will return to the clinic on Day 14 (or at time of early termination) for an end-of-study evaluation. Safety and tolerability assessments will be made on Days 7 and 14. Tolerability will be evaluated by subject-reported adverse events (AEs), nasal examinations, and vital signs assessments

ELIGIBILITY:
Inclusion Criteria:

1. Male/female subjects 12 years of age and older
2. Provide written informed consent/pediatric assent.
3. Subjects must have moderate-to-severe rhinitis, with one or more of the following present:

   1. Sleep disturbance
   2. Impairment of daily activities, leisure and/or sport
   3. Impairment of school or work
   4. Troublesome symptoms
4. Screening Visit: Have a 12-hour reflective TNSS of at least 8 out of a possible 12 and a congestion score of 2 or 3 on Visit 1
5. Randomization Visit: For the 3 days prior to Randomization and on the morning of Randomization, the sum of the 7 consecutive reflective AM and PM TNSS assessments shall be equal to or greater than 56, with a nasal congestion score equal to or greater than 14
6. Randomization Visit: instantaneous TNSS score of at least 8 and a congestion score of at least 2 just prior to beginning the onset of action assessment
7. Have taken at least 10 doses of the lead-in medication
8. Willing and able to comply with the study requirements
9. At least a 2-year history of SAR during the current allergy season
10. The presence of IgE-mediated hypersensitivity to a prevailing, individual, seasonal pollen, confirmed by a positive response to skin prick within the last year.
11. General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results.
12. Subjects receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit
13. Subjects currently receiving sublingual immunotherapy are excluded. A 6-month washout period is required following the last dose of sublingual immunotherapy.

Exclusion Criteria:

1. On Focused Nasal Examination, the presence of any superficial and moderate nasal mucosal erosion, nasal mucosal ulceration, or nasal septum perforation (Grade 1b - 4) at either the screening visit or randomization visit will disqualify the subject from the study.
2. Other nasal disease(s) likely to affect deposition of intranasal medication.
3. Nasal surgery or sinus surgery within the previous year.
4. Chronic sinusitis - more than 3 episodes per year
5. Planned travel outside of the pollen area during the study period
6. The use of any investigational drug within 30 days prior to Visit 1. No investigational products are permitted for use during the conduct of this study
7. Presence of any hypersensitivity to drugs similar to azelastine hydrochloride or fluticasone propionate
8. Women who are pregnant or nursing
9. Women of childbearing potential who are not abstinent or not practicing a medically acceptable method of contraception* see section 6.1.1
10. Respiratory Tract Infections within 14 days prior to Visit 1
11. Respiratory Tract Infections requiring antibiotic treatment 14 days prior to Visit 1
12. Asthma (with the exception of intermittent asthma).
13. Significant pulmonary disease including COPD
14. Clinically significant arrhythmia or symptomatic cardiac conditions
15. A known history of alcohol or drug abuse within the last 2 years
16. Existence of any surgical or medical condition or physical or laboratory findings, might significantly alter the absorption, distribution, metabolism, or excretion of study drug; that might significantly affect the subject's ability to complete this trial; or their safety in this trial.
17. Patients with a history of glaucoma
18. Clinically relevant abnormal physical findings within 1 week of randomization may preclude compliance with the study procedures
19. Employees of the research center or private practice and their family members
20. no more than 50% of their subjects have participated in protocol MP4001, MP4002 or MP4004

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1791 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (45):
- United States (45):
  - Allergy, Asthma and Immunology Associates, Scottsdale, Arizona
  - Clinical Research Center, Encinitas, California
  - AABI Associates Medical Group, Fountain Valley, California
  - Allergy & Asthma Care Center of So. Cal, Long Beach, California
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Allergy Associates Medical Group Inc, San Diego, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Bensch Research Associates, Stockton, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - Asthma and Allergy Associates, Colorado Springs, Colorado
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - Clinical Research Atlanta, Atlanta, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - Family Allergy and Asthma Reserach, Louisville, Kentucky
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Reseacrh Institute, Minneapolis, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - The Asthma and Allergy Center, Papillion, Nebraska
  - Atlantic Research Center, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Research Asthma, Sinus and Allergy Centers, Warren Township, New Jersey
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy and Consultants of NJ/PA, Collegeville, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy, Asthma and Urticaria of Charleston, Charleston, South Carolina
  - East Tennesse Center for Clinical Research, Knoxville, Tennessee
  - Allergy and Asthma Associates, Austin, Texas
  - Allergy and Asthma Center of Austin, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Pharmaceutical Research & Consulting Inc, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Diagnostic Research Group, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy, Asthma Research Center, San Antonio, Texas
  - Allergy and Asthma Center, Waco, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Intermountain Clinical Research, Draper, Utah
  - Asthma, Inc., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- MP29-02: azelastine HCl 548mcg / fluticasone propionate 200mcg
- Azelastine Hcl: azelastine HCl nasal spray
- Fluticasone Propionate: fluticasone propionate nasal spray
- Placebo: placebo nasal spray
Period: Overall Study
Arm/Group | MP29-02 | Azelastine Hcl | Fluticasone Propionate | Placebo
Started | 448 | 445 | 450 | 448
Completed | 434 | 430 | 431 | 433
Not Completed | 14 | 15 | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP29-02 | Azelastine Hcl | Fluticasone Propionate | Placebo | Total
Number analyzed (Participants) | 448 | 445 | 450 | 448 | 1791
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 38 | 56 | 46 | 197
  Between 18 and 65 years | 382 | 390 | 390 | 387 | 1549
  >=65 years | 9 | 17 | 4 | 15 | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 35.6 (14.5) | 36.4 (14.8) | 34.2 (14.5) | 34.7 (14.1) | 35.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 271 | 280 | 269 | 1097
  Male | 171 | 174 | 170 | 179 | 694
Region of Enrollment [Number; unit: participants]
  United States | 448 | 445 | 450 | 448 | 1791

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12 Hour Reflective Total Nasal Symptom Score (rTNSS)
Description: change from baseline in 12-hour reflective total nasal symptom score (rTNSS)consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary cards for the entire 14 day study period.The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.An greater negative value is suggestive of improvement.
Time Frame: day 1 to day 14
Population: Intent to Treat (ITT) population includes all subjects who had at least one post baseline dose efficacy evaluation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Azelastine Hcl | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 448 | 445 | 450 | 448
units on a scale | -5.5 (5.2) | -4.8 (4.8) | -4.9 (4.7) | -3.4 (4.3)

2. Secondary Outcome: Change From Baseline in 12 Hour Instantaneous Total Nasal Symptom Score (iTNSS)
Description: change from baseline in 12-hour instantaneous total nasal symptom score (iTNSS)consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary cards for the entire 14 day study period.The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.A greater negative score is suggestive of improved condition.
Time Frame: day 1 to day 14
Population: Intent to Treat (ITT) population includes all subjects who received at least one post baseline efficacy evaluation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Azelastine Hcl | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 448 | 443 | 450 | 448
units on a scale | -5.0 (5.3) | -4.3 (4.9) | -4.7 (4.9) | -3.1 (4.4)

3. Secondary Outcome: Change From Baseline in Adult Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Description: adult Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scored at day 1(baseline) and at day 14.The scale is measured from a value of 0 to 24. A negative number corresponds to a change from baseline measurement. An increased negative number is suggestive of improvement.
Time Frame: day 1 to day 14
Population: Intent to treat (ITT)population includes all subjects(18 years or older) who had at least one post baseline efficacy evaluation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Azelastine Hcl | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 381 | 394 | 384 | 393
units on a scale | -1.6 (1.3) | -1.4 (1.3) | -1.6 (1.2) | -1.0 (1.2)

ADVERSE EVENTS:
Arm/Group | MP29-02 | Azelastine Hcl | Fluticasone Propionate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/448 | 0/449 | 0/450 | 1/451
Other Adverse Events (participants affected / at risk) | 57/448 | 47/449 | 32/450 | 26/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP29-02 (N=448) | Azelastine Hcl (N=449) | Fluticasone Propionate (N=450) | Placebo (N=451)
lacerated right hand (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pyogenic arthritis right elbow (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP29-02 (N=448) | Azelastine Hcl (N=449) | Fluticasone Propionate (N=450) | Placebo (N=451)
dysgusia (Gastrointestinal disorders) | 21 (21) | 23 (23) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 10 (10) | 14 (14) | 8 (8) | 4 (4)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6) | 6 (6) | 8 (8)
oropharyngial pain (General disorders) | 5 (5) | 2 (2) | 6 (6) | 2 (2)
somnolence (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 5 (5)
mucosal erosion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators participating in multicenter studies must agree not to present data gathered individually or by a subgroup of centers before the full, initial publication, unless this has been agreed to by all other investigators and Meda Pharmaceuticals.

Meda Pharmaceuticals requests that it receive copies of any intended communication reasonably in advance (at least 15 working days for an abstract or oral presentation and 45 working days for a manuscript)